CLINICAL TRIAL: NCT04605562
Title: Precision Treatment of Locoregionally Advanced Nasopharyngeal Carcinoma Based on Molecular Immune Subtyping: an Umbrella Trial
Brief Title: Umbrella Biomarker-Guided Therapy in NPC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jun Ma, MD, Prof, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SZR2019-069
Record Dates: First submitted 2020-10-22; First posted 2020-10-28 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — palbociclib; Radiotherapy, Intensity-Modulated; LY-2157299

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IC+CCRT with palbociclib (Experimental): If patients were non-Immune Subtype.
  Interventions: Drug: GP+DDP; Drug: Palbociclib; Radiation: Intensity-modulated radiotherapy
- IC+CCRT with galunisertib and PD-1 blocking antibody (Experimental): If patients were Evaded Immune Subtype.
  Interventions: Drug: GP+DDP; Radiation: Intensity-modulated radiotherapy; Drug: PD-1 blocking antibody; Drug: Galunisertib
- IC+CCRT with PD-1 blocking antibody (Experimental): If patients were Active Immune Subtype.
  Interventions: Drug: GP+DDP; Radiation: Intensity-modulated radiotherapy; Drug: PD-1 blocking antibody

INTERVENTIONS:
Drug: GP+DDP — Gemcitabine as induction chemotherapy, 1000 mg/m2 day 1, 8 per cycle, every 3 weeks for 3 cycles; induction cisplatin 80mg/m2, every 3 weeks for 3 cycles before radiation; concurrent cisplatin 100mg/m2, every 3 weeks for 2 cycles during radiation
Drug: Palbociclib — Administered orally
  Arms: IC+CCRT with palbociclib
Radiation: Intensity-modulated radiotherapy — Definitive IMRT of 70 Gy, 33 fractions, 5 fractions/week, 1 fraction/day
Drug: PD-1 blocking antibody — Administered every 3 weeks
  Arms: IC+CCRT with PD-1 blocking antibody; IC+CCRT with galunisertib and PD-1 blocking antibody
Drug: Galunisertib — Administered orally
  Arms: IC+CCRT with galunisertib and PD-1 blocking antibody

SUMMARY:
This is a phase 2, open-label, umbrella study, with the purpose to evaluate the therapeutic efficacy and safety of chemoradiotherapy in combination with immunotherapy and/or targeted treatment in high-risk locoregionally advanced nasopharyngeal carcinoma. The specific grouping of patients' depends on the SYSUCC immune subtyping based on 100+ gene panel testing.

DETAILED DESCRIPTION:
This is a phase 2, open-label, umbrella study, with the purpose to evaluate the therapeutic efficacy and safety of chemoradiotherapy in combination with immunotherapy and/or targeted treatment in high-risk locoregionally advanced nasopharyngeal carcinoma. The specific grouping of patients' depends on the SYSUCC immune subtyping based on 100+ gene panel testing. The molecular subgroups include the Active, Evaded and non-Immune Subtypes. New treatment arms may be added and/or existing treatment arms may be closed during the study course on the basis of ongoing efficacy and safety as well as the current treatments available.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 65;
2. Pathological type: non-keratinizing carcinoma (World Health Organization criteria);
3. Diagnosed with LANPC (T4N1, T1-4N2-3) according to the 8th edition clinical staging system of the American Joint Committee on Cancer [AJCC]/Union for International Cancer Control [UICC];
4. ECOG performance score: 0 to 1;
5. Normal bone marrow function: white blood cell count > 4×109/L, hemoglobin > 90g/L, platelet count > 100×109/L;
6. Normal values of thyroid function, amylase and lipase examination, pituitary function, inflammation and infection indicators, myocardial enzymes, and ECG results. For patients older than 50 years with a smoking history, normal lung function are required. Patients with abnormal ECG and/or a history of vascular disease (but not meeting the exclusion criteria listed in the exclusion criteria 7) need further testing and require normal results of myocardial function and color Doppler ultrasound.
7. Normal liver and kidney function: total bilirubin ≤ 1.5 × upper limit of normal (ULN); alanine transaminase and aspartate transaminase ≤ 2.5 × ULN; alkaline phosphatase ≤ 2.5 × ULN; creatinine clearance rate ≥ 60 ml/min;
8. Patients must sign informed consent and be willing and able to comply with the requirements of visits, treatment, laboratory tests and other research requirements stipulated in the research schedule;
9. Subjects with pregnancy ability must agree to use reliable contraceptive measures from screening to 1 year after treatment.

Exclusion Criteria:

1. Hepatitis B virus surface antigen (HBsAg) positive and HBV DNA > 1×10E3 copies/ml; anti-hepatitis C virus positive;
2. Anti-human immunodeficiency virus (HIV) positive or diagnosed with acquired immune deficiency syndrome (AIDS);
3. Active tuberculosis: active tuberculosis in the past 1 year should be excluded regardless with treatment; history of active tuberculosis over 1 year should be excluded except that previous regulatory anti-tuberculosis treatment is proved;
4. Active, known or suspected autoimmune disease (including but not limited to uveitis, enteritis, hepatitis, pituitary, nephritis, vasculitis, hyperthyroidism, hypothyroidism and asthma requiring bronchiectasis). Exceptions are type I diabetes mellitus, hypothyroidism requiring hormone replacement therapy, skin disorders requiring no systemic treatment (such as vitiligo, psoriasis or alopecia);
5. Previous interstitial lung disease or pneumonia requiring oral or intravenous steroid therapy;
6. Chronic treatment with systemic glucocorticoid (dose equivalent to or over 10 mg prednisone per day) or any other form of immunosuppressive therapy. Subjects who used inhaled or topical corticosteroids were eligible;
7. Uncontrolled heart disease, for example: 1) heart failure (NYHA level ≥ 2); 2) unstable angina; 3) myocardial infarction in past 1 year; 4) supraventricular or ventricular arrhythmia requiring treatment or intervention;
8. Pregnant or lactating women (pregnancy test should be considered for women with sexual life and fertility);
9. Previous or concurrent with other malignant tumors, except for adequately treated non-melanoma skin cancer, cervical carcinoma in situ and thyroid papillary cancer;
10. Allergy to macromolecular protein preparations, or any component of the intervention drugs;
11. Active infection requiring systemic treatment;
12. History of organ transplantation;
13. History of psychotropic disease, alcoholism or drug abuse; other situation assessed by the investigators that may compromise the safety or compliance of patients, such as serious disease requiring timely treatment (including mental illness), severe laboratory abnormalities, or family-social risk factors.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival (FFS) | 3-year
  Failure-free survival is measured from day of diagnosis until treatment failure, death from any cause, or last follow-up visit, whichever occurred first

SECONDARY OUTCOMES:
Overall survival (OS) | 3-year
  Overall survival is measured from day of diagnosis until death due to any cause or the latest known date alive
Distant failure-free survival (DFFS) | 3-year
  Distant failure-free survival is measured from day of diagnosis until distant metastasis
Incidence rate of investigator-reported adverse events (AEs) | 3-year
  Analysis of investigator-reported adverse events (AEs) are based on treatment-related AEs (trAEs) and immune-related AEs (irAEs), and all-grade AEs and grade 3-4 AEs. AEs are evaluated by investigators according to the Common Terminology Criteria for Adverse Events, version 5.0
Incidence rate of patient-reported adverse events (AEs) | 3-year
  Analysis of patient-reported adverse events (AEs) are based on treatment-related AEs (trAEs) and immune-related AEs (irAEs), and all-grade AEs and grade 3-4 AEs. AEs are evaluated by patients themselves

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No